CLINICAL TRIAL: NCT05807542
Title: Prediction for pCR After Neoadjuvant Immunotherapy Combined With Chemotherapy Using Single-Cell RNA Sequencing in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma (ESCC) : A Single-Arm Phase II Clinical Trial
Brief Title: Neoadjuvant Immunotherapy Combined With Chemotherapy in Patients With Locally Advanced ESCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEEK-01
Record Dates: First submitted 2023-03-27; First posted 2023-04-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-03

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab combined with chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel-albumin; Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab will be administered on day 1 of each cycle at 200mg once every 21 days.
Drug: Paclitaxel-albumin — Paclitaxel-albumin will be administered on day 1 of each cycle at 260mg/m2 once every 21 days.
Drug: Carboplatin — carboplatin will be administered on day 1 of each cycle at AUC=5 once every 21 days.

SUMMARY:
Prediction for pCR After Neoadjuvant Immunotherapy Combined With Chemotherapy Using Single-Cell RNA Sequencing in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years ;
* Initially diagnosed patients with stage T2-4aN0-1M0 esophageal squamous cell carcinoma;
* No chemotherapy or any other antitumor therapy was used before inclusion
* ECOG score 0-1;
* Life expectancy is greater than 3 months;
* The patient has no indication for emergency surgery；
* No immediate childbearing requirement；
* The main organs function well, and the examination indicators meet the following requirements:

  i. Blood routine examination:
  1. Hemoglobin ≥90 g/L (no blood transfusion within 14 days);
  2. Neutrophil count ≥1.5×109/L;
  3. Platelet count ≥75×109/L; ii. Biochemical examination: iii. Total bilirubin ≤1.5×ULN (upper limit of normal); iv. Serum alanine aminotransferase (ALT) or serum alanine oxalacetic aminotransferase (AST) ≤ 2.5×ULN; v. Endogenous creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula);
* Sign informed consent;
* The compliance was good, and the family members agreed to cooperate with the survival follow-up.

Exclusion Criteria:

* Pregnant or nursing women；
* Patients with a history of other malignant diseases in the last 5 years, except cured skin cancer and cervical carcinoma in situ；
* Patients with a history of uncontrolled epilepsy, central nervous system disease or mental disorder whose clinical severity, as determined by the investigator, may prevent the signing of informed consent or affect the patient's adherence to medication use；
* Severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases；
* Allergic to any investigational drug ingredient；
* Any bleeding event with a severe grade of 3 or above CTCAE4.0 occurring within 4 weeks prior to screening;
* Patients with hypertension (systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg) who are not well controlled by single antihypertensive medication;History of unstable angina pectoris;Patients with newly diagnosed angina pectoris or myocardial infarction within 3 months prior to screening;Arrhythmias (including QTcF: male ≥450 ms) requiring long-term use of antiarrhythmic drugs and New York Heart Association grade ≥II cardiac insufficiency;
* Long-term unhealed wounds or incomplete healing fractures;
* Previous history of organ transplantation;
* Imaging shows that the tumor has invaded important blood vessels, or the investigator determines that the patient's tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during treatment;
* Patients with abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L) and bleeding tendency (14 days before randomization must meet the requirement that INR is within the normal range without the use of anticoagulants);Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogities;Low doses of warfarin (1 mg orally, once daily) or low doses of aspirin (up to 100 mg daily) are permitted for prophylactic purposes if INR ≤ 1.5;
* Occurrence of arteriovenous thrombosis within one year prior to screening, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis (except venous thrombosis caused by intravenous catheterization during previous chemotherapy and determined to be cured by researchers), pulmonary embolism, etc.;
* Those who have a history of psychotropic substance abuse and cannot abstain or have mental disorders;
* A history of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* In the investigator's judgment, there is a serious concomitant disease that endangers the patient's safety or interferes with the patient's completion of the study.
* Patients who did not meet the inclusion criteria, or who were considered unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Pathological complete response | 4 weeks after surgery
  Total tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Major pathological response | 4 weeks after surgery
  Total/moderate tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell
Objective Response Rate (ORR) | At the end of Cycle 3 (each cycle is 21 days)
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor

CONTACTS AND LOCATIONS:
Locations (1):
- ShanghaiZhongshan, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No